CLINICAL TRIAL: NCT06734793
Title: Pilot Study of Wearable Electronic Breath Sound Sensing Device for Monitoring of Breath Sounds in Pediatric Patients with Asthma
Brief Title: Wearable Electronic Breath Sound Sensing Device
Acronym: WEBSS
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other); Imlay Foundation (Unknown)
Responsible Party: Principal Investigator, Lokesh Guglani, Associate Professor, Emory University
Other Study IDs: STUDY00007232
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Asthma in Children; Asthma Attack
Keywords: Hospital admission; Wearable stethoscope; Asthma Exacerbations
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Pediatric patients with asthma: The study participants will be asked to wear up to a total of 5 patches in the following locations: left upper chest for the left upper lobe, left lower back for left lower lobe, right upper chest for the right upper lobe, right middle chest for the right middle lobe, and right lower back for the right lower lobe of the lung.
  Interventions: Device: Wearable stethoscope; Other: Routine Clinical lung Auscultation

INTERVENTIONS:
Device: Wearable stethoscope — The device is a soft, wearable stethoscope designed for continuous, comfortable monitoring of patients for abnormal breath sounds, such as wheezing, which can indicate asthma exacerbations. It automatically detects and diagnoses abnormal breath frequencies, wirelessly transmitting data for analysis. Preliminary materials have shown biocompatibility, ensuring the device is safe for use in children. A key feature is its machine-learning algorithm, which can classify and differentiate normal from abnormal sounds with an expected accuracy above 80%. Initial in vivo tests will compare the device's findings to those of a commercial-grade stethoscope in healthy subjects and individuals with asthma. Breath sound data will be used to improve the detection of wheezing sounds from these continuous recordings based on frequency and amplitude analysis of the recordings.
Other: Routine Clinical lung Auscultation — The study PI will auscultate the participant's lungs at enrollment to ensure that wheezing is present before beginning the continuous recording of the participant's lung sounds. The PI will assess the participant's respiratory status daily at the start of each breath sound recording session.
  Other Names: Standard of Care

SUMMARY:
This study will assess the ability of a wearable stethoscope to monitor wheezing in high-risk asthma patients admitted at Children's Healthcare of Atlanta.

This study is important to assist in the health management of patients with chronic lung diseases that can experience exacerbations leading to their health worsening and requiring hospitalization. The population that will be approached for this study will include 10 pediatric subjects hospitalized at Children's Healthcare of Atlanta for an asthma-related exacerbation. Participants will wear the patches for up to 8 hours on their chest and back wall from their date of consent until their hospital discharge. This may range from the participant taking part in 1 to 14 visits that could last up to 8 hours.

DETAILED DESCRIPTION:
The main goal of this study is to evaluate the ability of a novel wearable breath sound sensor (wearable stethoscope) to continuously monitor breath sounds, specifically wheezing, in pediatric asthma patients during hospital admission. The data collected will be used to develop a wheeze detection algorithm. The breath sound recordings from this device will not be used for any medical decision-making or treatment changes, and all study participants will continue to receive routine medical management per standard of care guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17 years
* Diagnosis of persistent asthma
* Being treated for an acute asthma exacerbation
* Parent can speak and understand English

Exclusion Criteria:

* Unable to provide consent for the study
* History of prematurity
* History of other chronic lung conditions - cystic fibrosis, bronchiectasis, or primary ciliary dyskinesia
* History of latex allergy or allergy to medical tape adhesive
* Patients currently using another medical device - implanted pacemaker or vagal nerve stimulator or diaphragm pacing device

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with asthma between the ages of 6-17 years who are being treated for an acute asthma exacerbation in the hospital.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Respiratory Score (CRS) change | Star of each recording session, end of each recording session up to 14 days
  CRS is a 12-point assessment used to evaluate respiratory distress in hospitalized patients and guide treatment for asthma and bronchiolitis. It measures factors such as respiratory rate, work of breathing, wheezing, hypoxia, dyspnea, and cough. The change in CRS score will be recorded at the beginning and end of each session and later correlated with changes in breath sound recordings from the device. The absolute change in CRS will be correlated with changes in the breath sound recordings.

SECONDARY OUTCOMES:
Detection of wheezing sounds by the wearable stethoscope | Throughout study participation until hospital discharge (up to 14 days)
  Detection of wheezing using convolutional neural networks and testing the wearable stethoscope's reliability against wheezing detected by medical providers during the participants' hospital stay until discharge up to 14 days.
Visual Erythema Assessment Scale (VEAS) | At the end of each recording session up until hospital discharge (up to 14 days)
  VEAS will be used to assess skin changes after the recording is completed. VEAS evaluates the degree of erythema (redness) on the skin, which is often an indicator of inflammation or irritation. The scoring is based on visual observation, focusing on the intensity and extent of redness, with scores ranging from 0 (no reaction) to 9 (most intense reaction). Higher scores indicate more severe redness or inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Lokesh Guglani, MD, Principal Investigator — Emory University
Locations (1):
- Arthur M. Blank Hospital | Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers will only share data published in aggregate as part of a manuscript or abstract.
Time Frame: Data will be published in the form of a peer-reviewed manuscript by the end of 2025.